CLINICAL TRIAL: NCT06848049
Title: Effect of Mobile Application-Assisted Nursing Services on Pressure Injury Management: A Randomized Controlled Trial on Patients Receiving Home Care
Brief Title: Mobile Application-Assisted Pressure Injury Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Rukiye Kokkiz, Lecturer, Fenerbahce University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 02.2025fbu
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pressure Injury; Nursing Caries; Application Site Wound
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Aplication (Experimental)
  Interventions: Other: Mobile Aplication
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Mobile Aplication — In this study, individuals will be monitored for 28 days. They will be asked to fill out the Pressure Injury Information Form and the Pressure Injury Skills Checklist for Caregivers to be informed about pressures throughout the study process. The researcher will fill out the Bates-Jensen Wound Assessment Tool to ensure that their pressures are improving. Individuals who will undergo the intervention will use the mobile application. Face-to-face training will be provided to individuals. Individual-specific audio reminders will be based on daily living activities and will be delivered via the mobile application according to changes in individual dependencies. After 30 days, individuals will be asked to fill out the Mobile Health Application Acceptance Scale, the Pressure Injury Knowledge Scale for Caregivers, and the Pressure Injury Skills Checklist. The Bates-Jensen Wound Assessment Tool will be filled out by the researcher.
  Arms: Mobile Aplication
Other: Control — In this study, individuals will be monitored for 28 days. In order to monitor their knowledge about pressure injuries, individuals will be asked to complete the Pressure Injury Information Form for Caregivers and the Pressure Injury Skills Checklist to monitor their skill levels about pressure injuries throughout the study period. The Bates-Jensen Wound Assessment Tool will be completed by the researcher to perform a physical examination of the patient and to assess the healing of the individual's pressure injury. Individuals in the control group will be interviewed twice by phone. Individuals with pressure injuries will be trained by a team consisting of a physician, nurse, dietician, and physiotherapist. Individuals will be interviewed twice by phone. After 30 days, individuals will be asked to complete the Mobile Health Application Acceptance Scale, the Pressure Injury Knowledge Scale for Caregivers, and the Pressure Injury Skills Checklist.
  Arms: Control

SUMMARY:
Pressure injuries develop due to decreased movement, especially in bedridden individuals receiving home care. In Turkey, the management of pressure injuries is carried out by nurses in acute and long-term care settings, and mostly by caregivers for individuals receiving home care. Studies have shown that individuals providing home care have a significant need for training. Today, digital health technologies are used to facilitate access to healthcare professionals and provide workload and cost efficiency. Telehealth services in these technologies can be provided via telephone or mobile applications. In this context, the aim of the study is to examine the effect of nursing services provided via mobile applications on the management of pressure injuries in individuals receiving home care. The study was designed as a randomized controlled experimental type. In the power analysis conducted to calculate the sample size, the sample size was determined as 56, and considering that there may be data losses, 60 people will be included in the study. The "Structured Information Form, Pressure Injury Information Form for Caregivers, Pressure Injury Skill Checklist for Caregivers, and Pressure Injury Follow-up Form" will be used as data collection tools in the study. In this study, it is thought that the nurse's remote monitoring of individuals receiving home care with a mobile application in the management of pressure injuries will contribute to patient safety and care costs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals receiving home care and caregivers
* Individuals over the age of 18
* Individuals with a caregiver who can use the mobile application (The mobile application will be introduced to the caregivers in the first meeting and consent will be obtained from the individual to use it)
* Individuals with a smartphone
* Individuals who can use a smartphone
* Individuals who fill in the data completely
* Individuals with a pressure injury

Exclusion Criteria:

* Individuals who cannot use mobile applications
* Individuals who cannot use smartphones
* Individuals who want to leave the study
* Individuals who have incomplete data collected in the study for various reasons
* Individuals with chronic diseases (Diabetes and Hypertension)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Improvement (decrease) in the Bates-Jensen Wound Assessment Tool scores of individuals receiving nursing services will be observed with the mobile application developed for the management of pressure injuries. | 28 days
  The assessment tool developed by Bates-Jensen et al. in 1992 is a scale that broadly addresses the physiological and anatomical characteristics of the wound. It consists of 13 items: size, depth, edges, tunneling, type and amount of necrotic tissue, type and amount of exudate, color of the skin around the wound, peripheral tissue edema and induration, granulation tissue and epithelialization. As a result of the scale scoring, 1 point indicates that the wound is in better condition, while 5 points indicate that the wound condition is worse. In the presence of necrotic tissue, the type and amount of necrosis are also included in the assessment. The total score obtained varies between 13-65, and an increase in the score indicates that the wound condition is worsening.
Improvement (increase) will be observed in the "Pressure Injury Knowledge Scale for Caregivers" scores of caregivers receiving nursing services through the mobile application developed for the management of pressure injuries. | 28 days
  The Pressure Injury Patient Information Form was prepared by the researcher in line with the literature. There are questions about the management of pressure injuries. The form consists of 15 questions. Each question is 1 point, the lowest score is "0" and the highest score is "15". As the score increases, the knowledge of individuals to manage pressure injuries increases. Before starting the research, expert opinions will be presented and arrangements will be made.
Improvement (increase) will be observed in the "Pressure Injury Skills Checklist" scores of caregivers receiving nursing services through the mobile application developed for the management of pressure injuries. | 28 days
  The Pressure Injury Skill Form was prepared by the researcher in line with the literature. The form consists of 10 items. For each item, "Not Applied" was evaluated as "0" points, "Partially Applied" as "1" points, and "Applied" as "2" points. The lowest score to be received from the checklist is "0" and the highest score is "20". An increase in the score indicates that the individual's pressure injury skills have improved. Before starting the research, it will be presented to expert opinions and arrangements will be made.